CLINICAL TRIAL: NCT00661856
Title: The Effect of Increased Soy Protein Intake on Bone Metabolism
Brief Title: Effect of Soy Isoflavones on Bone Mineral Density and Physical Performance Indices
Acronym: SoyPTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Solae, LLC (Industry)
Responsible Party: J C Gallagher, Creighton University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0012254
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Osteoporosis
Keywords: Soy Isoflavones, Bone Mineral Density, Post menopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Soybean Proteins; Genistein; daidzein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Soy Protein group 25g of Soy protein with no Isoflavones
  Interventions: Dietary Supplement: Soy protein
- 2 (Experimental): Soy Isoflavone group 25g of Soy Protein with 90mg of Isoflavones
  Interventions: Dietary Supplement: Soy protein
- 3 (Placebo Comparator): 25g of Milk protein
  Interventions: Dietary Supplement: Soy protein

INTERVENTIONS:
Dietary Supplement: Soy protein — 25g of Soy protein with or with out 90mg of isoflavones ones a day given for a period of 24 months
  Other Names: genistein, daidzein, glycetein

SUMMARY:
The aim of the present study was to investigate the effects of soy and soy plus isoflavones on bone mineral Density and physical performance in post menopausal women.

DETAILED DESCRIPTION:
Post menopausal estrogen deficiency causes physiologic changes in body composition including decreased lean body weight and bone mass. A decrease in muscle strength along with osteoporosis puts post menopausal women at a high risk of hip fractures causing considerable mortality and morbidity. Estrogen use has been shown to reduce bone density loss and increase muscle strength but given the concerns regarding its use, patients are looking for alternatives such as Soy isoflavones. Most human studies on the effect of Soy on bone mineral density (BMD) in post menopausal women have been short term i.e. 3-6 months and failed to provide conclusive evidence. There is no evidence of its effects on physical performance.

The aim of the present study is to investigate the effects of 25g of soy protein alone or with 90mg of isoflavones on bone mineral Density and physical performance indices in post menopausal women over a duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* at least 55-75 years of age
* at least 7 years post menopausal either spontaneous or surgical

Exclusion Criteria:

* must not have used estrogen for atleast 2 months prior to entering study
* must be on no bone active drugs such as bisphosphonates, anti convulsants, calcitonin and long term steroids
* osteoporosis (T-score<-2.5)
* BMI <18 or >34

Ages: 55 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2001-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 24 months

SECONDARY OUTCOMES:
Physical Performance Indices | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: J C Gallagher, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Gallagher JC, Satpathy R, Rafferty K, Haynatzka V. The effect of soy protein isolate on bone metabolism. Menopause. 2004 May-Jun;11(3):290-8. doi: 10.1097/01.gme.0000097845.95550.71. PMID 15167308